CLINICAL TRIAL: NCT04717453
Title: A Study to Characterize Rate of Ureagenesis Utilizing Oral [1-13C] Sodium Acetate in the Spectrum of Severity of Patients With Ornithine Transcarbamylase (OTC) Deficiency
Brief Title: Study to Characterize Rate of Ureagenesis in Patients With Ornithine Transcarbamylase (OTC) Deficiency
Status: Terminated | Type: Observational
Why Stopped: Sponsor's Decision
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: DTX301-CL102
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Ornithine Transcarbamylase Deficiency
Keywords: OTC; OTC Deficiency; Neonatal; Late Onset; Asymptomatic Carrier
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA for OTC genotype
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult Patients with OTC Deficiency: Eligible subjects will be asked to participate in 5 clinic visits, each lasting up to 3 days. Each visit will assess rate of ureagenesis during the 4 hours following ingestion of [1-13C]sodium acetate. Sodium acetate is used as a tracer to measure the rate of ureagenesis. Patient interview, reported outcomes and cognitive assessments will take place over the 3 days.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The objectives of the study are to characterize urea production rates in patients with OTC, characterize the association of rate of ureagenesis and disease severity in OTC patients, characterize the association of rate of ureagenesis and executive and verbal function and characterize the association of rate of ureagenesis and patient-reported functional status.

DETAILED DESCRIPTION:
Study DTX301-CL102 is a noninterventional, observational study to characterize the rate of ureagenesis and to assess neurocognition and functional status in the spectrum of OTC deficiency and their association with biochemical characteristics. [1-13C]Sodium acetate will be administered orally as a tracer to measure the rate of ureagenesis.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent.
* For symptomatic patients:
* Confirmed clinical diagnosis of OTC deficiency and enzymatic, biochemical, or molecular testing.
* Documented history of ≥ 1 symptomatic hyperammonemic episode with ammonia level ≥ 100 μmol/L
* Patients on ongoing daily ammonia scavenger therapy must be at a stable dose(s) for ≥ 4 weeks prior to Visit 1 (Baseline)
* For asymptomatic patients: confirmed diagnosis of OTC deficiency by family history and documented by molecular testing.
* Willing and able to comply with the study procedures and requirements, including clinic visits, blood and urine collections, questionnaires, and cognitive assessments.

Key Exclusion Criteria:

* Liver transplant, including hepatocyte cell therapy/transplant.
* History of liver disease
* Significant hepatic inflammation or cirrhosis
* Participation in another investigational medicine study within 3 months of Screening
* Participation (current or previous) in another gene transfer study
* Pregnant or nursing

Other protocol specific criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 30 patients will be enrolled, with up to 6 (20%) asymptomatic patients and at least 18 (60%) patients with late-onset OTC deficiency.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Rate over time of ureagenesis for 4 hours based on presence of [1-13C] in urea | Predose (0hour) up to 4 hours post dose at Baseline, Weeks 24, 48, 72, and 96
  Urea excretion after ingestion of sodium acetate as measured in blood
OTC Genotype | Up to 96 weeks
  Genotype in blood
Rate of Hyperammonemic Crisis (HAC) | Up to 96 weeks
Cognitive assessment | Up to 96 weeks
  Cogstate platform
Hyperammonemia Indicator Questionnaire (HI-Q) | Up to 96 weeks
  Patient-reported outcome (PRO) for symptoms of hyperammonemia
OTC Deficiency Impact Questionnaire (OTC-D-IQ) | Up to 96 weeks
  PRO for impact of hyperammonemia

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceuticals
Locations (1):
- PPD Phase 1 Clinic - Orlando, Orlando, Florida, United States